CLINICAL TRIAL: NCT03659266
Title: Effects of Combined Treatment by Botulinum Toxin A and Robot-Assisted Gait Training (Lokomat®) on Walking Ability in Patients With Chronic Stroke: a Prospective, Controlled, Randomized Study
Brief Title: Effects of Combined Treatment by Botulinum Toxin and Lokomat® on Walking Ability in Chronic Stroke
Acronym: Lokomat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017-69
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2022-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): D0: Injection of Botulinum toxin A in triceps surae, according to pre-established modalities (no influence of the experimental protocol on this stage) W2-W4: Robotic walking rehabilitation by Lokomat® in the functional rehabilitation department (conventional hospitalization) W4-W6: Return to home, "wash-out"period W6-W8: Conventional walking rehabilitation in the functional rehabilitation department (conventional hospitalization)
  Interventions: Other: Robotic walking rehabilitation by Lokomat®; Other: Conventional walking rehabilitation
- group 2 (Active Comparator): D0: Injection of Botulinum toxin A in triceps surae W2-W4: Conventional walking rehabilitation in the functional rehabilitation department (conventional hospitalization) W4-W6: Return to home, "wash-out"period W6-W8: Robotic walking rehabilitation by Lokomat® in the functional rehabilitation department (conventional hospitalization)
  Interventions: Other: Robotic walking rehabilitation by Lokomat®; Other: Conventional walking rehabilitation

INTERVENTIONS:
Other: Robotic walking rehabilitation by Lokomat® — Lokomat sessions / week for 2 weeks. Each session lasts 45 minutes including 30 minutes of effective work of the march and 15 minutes of setting up.
Other: Conventional walking rehabilitation — 5 physiotherapy sessions / week for 2 weeks. Each session lasts 45 minutes including 30 minutes of walking and 15 minutes of stretching

SUMMARY:
75% patients in the chronic phase of a stroke keep walking disabilities. Focal spasticity in the paretic lower limb frequently causes these walking disabilities, and the gold standard treatment is intramuscular injection of Botulinum toxin A in the spastic muscles.

To potentiate the effects of toxin, walking rehabilitation is usually prescribed in the weeks following injection, but the protocols vary and few have been evaluated in the medical literature.

In particular, the effect on walking ability of combined treatment by botulinum toxin A and robot-assisted gait training has never been evaluated.

Tested hypothesis: Robot-assisted gait training by Lokomat® motorized exoskeleton potentiates botulinum toxin's effects better than conventional walking therapy.

The aim of this study was to evaluate the effects on walking ability of the association of focal spasticity treatment by Botulinum toxin and Lokomat-assisted walking rehabilitation in patients suffering from spastic hemiparesia after stroke in the chronic phase.

Outcome:

-Primary: distance walked (meters) in the six-minute walk test (SMWT)

Prospective, randomized, controlled, opened, monocentric study with a crossover design.

Recruitment of patients over 18 years of age, in the chronic phase of stroke, who have already been treated by Botulinum toxin injection for focal spasticity in our PMR ward.

Assessment at Day one (D0), Week four (W4) and Week eight (W8).

Following a preliminary study which had the six-minute walk test as a secondary outcome, the expected results are a significant improvement of the distance walked in the SMWT after robotic rehabilitation, and a lack of significant improvement following conventional therapy.

The study should serve to further harmonize and optimize rehabilitation protocols after toxin injections, and to justify the use of robotic rehabilitation for patients in the chronic phase of stroke.

DETAILED DESCRIPTION:
Introduction :

75% patients in the chronic phase of a stroke (>6 months) keep walking disabilities. Focal spasticity in the paretic lower limb frequently causes these walking disabilities, and the gold standard treatment is intramuscular injection of Botulinum toxin A in the spastic muscles.

To potentiate the effects of toxin, walking rehabilitation is usually prescribed in the weeks following injection, but the protocols vary and few have been evaluated in the medical literature.

In particular, the effect on walking ability of combined treatment by botulinum toxin A and robot-assisted gait training has never been evaluated.

Materials and Methods:

Tested hypothesis:

Robot-assisted gait training by Lokomat® motorized exoskeleton potentiates botulinum toxin's effects better than conventional walking therapy.

Aims:

* Primary: to evaluate the effects on walking ability of the association of focal spasticity treatment by Botulinum toxin and Lokomat-assisted walking rehabilitation in patients suffering from spastic hemiparesia after stroke in the chronic phase.
* Secondary: to determine the optimal time between the toxin injection and the start of robotic rehabilitation; to evaluate the effects of the combined treatment on the balance and spasticity.

Outcome:

* Primary: distance walked (meters) in the six-minute walk test (SMWT)
* Secondary: walking speed (meters/seconds), balance (Timed Up and Go Test, Berg Balance Scale), spasticity (score on the Modified Ashworth Scale and joint range of motion)

Study Design:

Prospective, randomized, controlled, opened, monocentric study with a crossover design.

Recruitment of patients over 18 years of age, in the chronic phase of stroke, who have already been treated by Botulinum toxin injection for focal spasticity in our PMR ward.

Assessment at Day one (D0), Week four (W4) and Week eight (W8).

1. st Group D0: Injection of Botulinum toxin A in triceps surae, according to pre-established modalities (no influence of the experimental protocol on this stage) W2-W4: Robotic walking rehabilitation by Lokomat® in the functional rehabilitation department (conventional hospitalization) W4-W6: Return to home, "wash-out"period W6-W8: Conventional walking rehabilitation in the functional rehabilitation department (conventional hospitalization)
2. nd Group: D0: Injection of Botulinum toxin A in triceps surae W2-W4: Conventional walking rehabilitation in the functional rehabilitation department (conventional hospitalization) W4-W6: Return to home, "wash-out"period W6-W8: Robotic walking rehabilitation by Lokomat® in the functional rehabilitation department (conventional hospitalization)

Expected results:

Following a preliminary study which had the six-minute walk test as a secondary outcome, the expected results are a significant improvement of the distance walked in the SMWT after robotic rehabilitation, and a lack of significant improvement following conventional therapy.

The study should serve to further harmonize and optimize rehabilitation protocols after toxin injections, and to justify the use of robotic rehabilitation for patients in the chronic phase of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Left or right spastic hemiparesia after a single unilateral hemorrhagic or ischemic stroke, in chronic phase (at least 6 months after stroke)
* Functional hindrance in walking
* Spasticity of paretic triceps surae allowing for focal treatment by Botulinum toxin injection

Exclusion Criteria:

* Inability to walk with or without technical aids >5min
* Cognitive disorders disallowing informed consent
* Spasticity equal or superior to 4 on the triceps surae (On the Modified Ashworth Scale)
* Physical exercise not allowed: non stable cardiovascular or pulmonary disease in particular
* Lokomat® use not allowed: cutaneous lesions that could come in contact with the straps, non consolidated recent fracture (<3months), severe disability in controlling trunk balance disallowing correct posture in Lokomat®, intra-abdominal cranial flap, weight>135kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Time of Ten-meter walk test | 20 minutes
  Time is measure while the individual walks the set distance (10 meters). the distance covered is divided by the time it took the individual to walk that distance

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France